CLINICAL TRIAL: NCT04433676
Title: Risk of Early Postoperative Nausea and Vomiting (PONV) - a Study With Data From the Swedish Perioperative Register (SPOR).
Brief Title: Early PONV - a Registry Based Study in Sweden.
Acronym: SPOR-PONV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jakob Wallden (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor-Investigator, Jakob Wallden, Senior Lecturer, Consultant Anesthesiologist, Västernorrland County Council, Sweden
Organization: Västernorrland County Council, Sweden (Other Government)
Other Study IDs: SPOR-PONV 1.0
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Complications
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with surgical procedures: Adult patients undergoing surgical procedures under general or regional anesthesia and with an admission to a recovery unit for the initial postoperative care.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The study is an registry study based on data from the Swedish Perioperative Registry (SPOR) during the years 2016-2022 with the aim to explore the risk for postoperative nausea and vomiting at the recovery unit (early PONV). The study will explore several cohorts (for example a specific procedure) on a national basis, report the risk for early PONV and identify associated factors.

DETAILED DESCRIPTION:
The study is a registry study based on data from the Swedish Perioperative Registry (SPOR) during the years 2016-2022 with the aim to explore the risk for postoperative nausea and vomiting at the recovery unit (early PONV).

Almost all hospitals in Sweden report surgical procedures to SPOR and for the years 2016-2019 there are almost 1.7 million procedures in the registry for patients >18years. Data will be extracted from SPOR on a yearly basis and results will be reported on selected cohorts (time periods and/or type of surgical procedure) during the study period.

There is an option for hospitals to register nausea and vomiting occurring at the recovery unit and submit the data to SPOR. If a hospital choose to use the variable in their dataset, all patients at their unit needs to be registered either with [No_Nausea or Vomiting], [Nausea] or [Nausea or Vomiting]. In the year 2019, more than 50% of procedures under anesthesia in the registry had registration of PONV. The strength with this system is that if a unit uses the variable, all cases will be classified either as "noPONV" or "PONV".

The investigators aim to use the variable PONV at the recovery unit to describe the risk for early PONV and explore associated factors in several cohorts of surgical procedures in Sweden.

The first dataset (2016-2018) was sent to the investigators from the SPOR registry in May 2019 and during the period June 2019- May 2020, the dataset was used to build up a model for the analysis of data with a preliminary report of elective surgeries in Sweden the year 2017.

An updated dataset (all cases 2016-2019) was retrieved from SPOR on June 3 2020 and further analysis and reporting is based on the most updated dataset (yearly basis).

ELIGIBILITY:
Inclusion Criteria:

* Procedure under general or regional anaesthesia
* Age >=18 years at the day of the procedure.

Exclusion Criteria:

* No entry of the PONV-variable in the SPOR-registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry data of patients with surgical procedures under general or regional anesthesia in Sweden 2016-2022.
Sampling Method: Probability Sample
Enrollment: 1500000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
PONV | At the recovery unit, up to 24 hours after surgery.
  Nausea or Vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Wallden, MD PhD, Principal Investigator — Region Västernorrland (Västernorrland County Council)
Locations (1):
- Västernorrland County Council / Sundsvall Hospital, Sundsvall, X, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Our dataset includes a large set of registry data, and we are not sure if we legally are allowed to share these data.

REFERENCES:
- [Derived] Wallden J, Larsson M, Moraitis A, Ahlqvist S, Cengiz Y, Myrberg T, Nystrom H, Hultin M. Early Postoperative Nausea and Vomiting After Bariatric Surgery: A Study of 8426 Patients from the Swedish Perioperative Registry (SPOR). Obes Surg. 2025 Dec;35(12):5308-5315. doi: 10.1007/s11695-025-08351-0. Epub 2025 Nov 4. PMID 41188673